CLINICAL TRIAL: NCT06432309
Title: Efficacy and Safety of Opicapone in Parkinson's Disease Add -on to Levodopa Carbidopa Intestinal Gel
Brief Title: Opicapone as Adjunctive Therapy to Levodopa-Carbidopa Intestinal Gel in Parkinson's Disease
Acronym: OPAILEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 480/2022/Oss/AOUFe
Record Dates: First submitted 2024-05-07; First posted 2024-05-29 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease; Effect of Drug
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; carbidopa, levodopa drug combination; Levodopa

STUDY DESIGN:
Intervention Model Description: Prospective randomised blinded End-point study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nOPC: Duodopa (Levodopa/carbidopa intestinal gel) in monotherapy (Other): Levodopa carbidopa intestinal gel infusion. Diurnal infusion from 7.a.m to 11 p.m.
  Interventions: Drug: Duodopa
- add-OPC: Duodopa plus OPC therapy (Active Comparator): Levodopa carbidopa intestinal gel infusion (Diurnal infusion from 7 a.m to 11 p.m) plus Opicapone 50 mg 1 tablet at nighttime (11 p.m)
  Interventions: Drug: Opicapone 50 mg; Drug: Duodopa

INTERVENTIONS:
Drug: Opicapone 50 mg — Evaluate the addition of the COMT-I, Opicapone, to the Levodopa-Carbidopa intestinal gel in Parkinson's Disease patients with motor fluctuations.
  Other Names: OPC
  Arms: add-OPC: Duodopa plus OPC therapy
Drug: Duodopa — Evaluate Levodopa-Carbidopa intestinal gel in Parkinson's Disease patients with motor fluctuations.
  Other Names: Levodopa/carbidopa intestinal gel (LCIG)

SUMMARY:
Levodopa-Carbidopa intestinal gel (LCIG) is an effective therapy for complicated Parkinson's disease (PD). Few studies have explored the efficacy and safety of the potential combination of LCIG with catechol-O-methyltransferase (COMT) inhibitors, particularly Opicapone (OPC).

DETAILED DESCRIPTION:
22 PD patients were randomized into LCIG monotherapy (n-OPC 11 patients) and LCIG+OPC (add-OPC 11 patients), further divided according to OPC adding time (E-OPC within one month and L-OPC after one month from LCIG implant).

Data on PD clinical aspects, Montreal Cognitive Assessment (MoCA), Unified Parkinson's Disease Rating Scale (UPDRS), Unified Dyskinesia Rating Scale (UDysRS), electroneurography (ENG), and pharmacological therapy (Levodopa Equivalent Dose-LEDD) were collected before LCIG implanted (T0) and in the following 12 (T1) months.

ELIGIBILITY:
Inclusion Criteria:

1. LCIG implantation not longer than 30 months before the study enrollment,
2. Presence of nocturnal akinesia (assessed by medical history and through item 2.9 of MDS-UPDRS part II (> 2), or/and
3. Persistence of morning or afternoon akinesia (assessed by item 4.3 in MDS UPDRS -IV( >2 ).

Exclusion Criteria:

1. Hoehn & Yahr (H&Y) >4,
2. Cognitive decline (MOCA< 17),
3. more than 30 months after LCIG positioning,
4. not compliant with treatment and follow-up visits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of motor fluctuations changes | 12 months
  Changes in MDS-UPDRS part IV from the initial assessment to 12 months follow-up.
Evaluation of dyskinesia changes | 12 months
  Changes in UDysRS from the initial assessment to 12 months follow-up.

SECONDARY OUTCOMES:
Changes in non-motor aspects of patients' daily living experiences | 12 months
  Changes of MDS-UPDRS I score from the initial assessment to 12 months follow-up.
Changes in motor aspects of patients' daily living experiences | 12 months
  Changes of of MDS-UPDRS II score from the initial assessment to 12 months follow-up.
Changes in non-motor symptoms in Parkinson's disease-cognition | 12 months
  Changes of MOCA score from the initial assessment to 12 months follow-up.
Neurophysiological outcome | 12 months
  Changes of sural amplitude potential through electroneurography from the initial assessment to 12 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Mariachiara Sensi, MD-Phd, Principal Investigator — Azienda Ospedaliero -Universitaria S. Anna Ferrara
Locations (1):
- University Hospital of Ferrara - Arcispedale Sant'Anna, Ferrara, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nyholm D, Jost WH. Levodopa-entacapone-carbidopa intestinal gel infusion in advanced Parkinson's disease: real-world experience and practical guidance. Ther Adv Neurol Disord. 2022 Jun 26;15:17562864221108018. doi: 10.1177/17562864221108018. eCollection 2022. PMID 35785401
- [Background] Fabbri M, Ferreira JJ, Lees A, Stocchi F, Poewe W, Tolosa E, Rascol O. Opicapone for the treatment of Parkinson's disease: A review of a new licensed medicine. Mov Disord. 2018 Oct;33(10):1528-1539. doi: 10.1002/mds.27475. Epub 2018 Sep 27. PMID 30264443
- [Background] Ikenaka K, Kajiyama Y, Aguirre C, Choong CJ, Taniguchi S, Doi J, Wang N, Ajiki T, Ogawa K, Kakuda K, Kimura Y, Mochizuki H. Decreased hepatic enzymes reflect the decreased vitamin B6 levels in Parkinson's disease patients. Pharmacol Res Perspect. 2024 Feb;12(1):e1174. doi: 10.1002/prp2.1174. PMID 38287715
- [Result] Leta V, van Wamelen DJ, Sauerbier A, Jones S, Parry M, Rizos A, Chaudhuri KR. Opicapone and Levodopa-Carbidopa Intestinal Gel Infusion: The Way Forward Towards Cost Savings for Healthcare Systems? J Parkinsons Dis. 2020;10(4):1535-1539. doi: 10.3233/JPD-202022. PMID 32597817